CLINICAL TRIAL: NCT03139162
Title: Development of Frailty and Complexity Indices From Data Collected With Resident Assessment Instrument - Home Care Adapted for Switzerland
Brief Title: Development of Clinical Indicators From the Swiss RAI-HC
Acronym: IndiRAI
Status: Completed | Type: Observational
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: Institution genevoise de maintien à domicile (Unknown)
Responsible Party: Principal Investigator, Catherine Ludwig, Professor, School of Health Sciences Geneva
Other Study IDs: 74217
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-10

CONDITIONS: Frail Elderly Syndrome
Keywords: Home Care Services; Aging; Frailty; Complexity; Nursing
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Swiss RAI-HC assessment — RAI-HC assessments done by trained nurses in clinical routine

SUMMARY:
The project aims at deriving frailty (FI) and complexity (CI) indices from data collected with the Resident Instrument Assessment - Home Care adapted for Switzerland (RAI-HC). Data were collected in 2015 by trained nurses in clinical routine with the primary purposes of health state assessment and individual home care planning. The study consists in a retrospective secondary analysis of health data from the Minimal Data Set (MDS), used to derive frailty and complexity indices according to published definitions and guidelines for index derivation. The analysis further aims at estimating the predictive power of these indices on undesirable health outcomes (falls, hospitalizations and deaths). The goal is to provide home care institutions and nurses valid algorithms to compute useful clinical indicators without additional assessment that the one routinely done with the RAI-HC.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older who were assessed in 2015 with the Swiss RAI-HC in clinical routine for care planning by the Geneva Institution for Home care and Assistance (imad) in Geneva, Switzerland

Exclusion Criteria:

* Men and women aged 17 or younger and/or who did not receive a full RAI-HC assessment in 2015

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult applicants for home care services provided by imad (Geneva, Switzerland) who received a first RAI-HC assessment in 2015 for routine care planning purposes
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Frailty Index | 1 year
  Index with a value ranging from 0 to 100, computed as the sum of health deficits recorded with the RAI-HC MDS divided by the number of deficits considered
Complexity Index | 1 year
  Index with a value ranging from 0 to 100, computed as the sum of complexity items recorded with the RAI-HC MDS divided by the number of items considered

SECONDARY OUTCOMES:
Falls | 6 months on average
  Falls recorded by means of follow-up RAI-HC assessments
Hospitalizations | 6 months on average
  Hospitalizations recorded by means of follow-up RAI-HC assessments
Mortality | through study completion, an average of 5 year
  Deceased (yes/no); collected through administrative records

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Ludwig, PhD, Principal Investigator — School of Health Sciences Geneva

IPD SHARING:
Plan to Share IPD: No
The coded datasets supporting the findings of this study are not publicly available for they belong to imad and are not the property of the authors of the study. The data analyzed for the study could be made available from the authors upon reasonable request and with prior agreement by imad.

REFERENCES:
- [Background] Hubbard RE, Peel NM, Samanta M, Gray LC, Fries BE, Mitnitski A, Rockwood K. Derivation of a frailty index from the interRAI acute care instrument. BMC Geriatr. 2015 Mar 18;15:27. doi: 10.1186/s12877-015-0026-z. PMID 25887105
- [Background] Loeb DF, Binswanger IA, Candrian C, Bayliss EA. Primary care physician insights into a typology of the complex patient in primary care. Ann Fam Med. 2015 Sep;13(5):451-5. doi: 10.1370/afm.1840. PMID 26371266
- [Background] Morris JN, Fries BE, Steel K, Ikegami N, Bernabei R, Carpenter GI, Gilgen R, Hirdes JP, Topinkova E. Comprehensive clinical assessment in community setting: applicability of the MDS-HC. J Am Geriatr Soc. 1997 Aug;45(8):1017-24. doi: 10.1111/j.1532-5415.1997.tb02975.x. PMID 9256857
- [Background] Armstrong JJ, Stolee P, Hirdes JP, Poss JW. Examining three frailty conceptualizations in their ability to predict negative outcomes for home-care clients. Age Ageing. 2010 Nov;39(6):755-8. doi: 10.1093/ageing/afq121. Epub 2010 Sep 21. No abstract available. PMID 20858672
- [Derived] Ludwig C, Busnel C. Derivation of a frailty index from the resident assessment instrument - home care adapted for Switzerland: a study based on retrospective data analysis. BMC Geriatr. 2017 Sep 7;17(1):205. doi: 10.1186/s12877-017-0604-3. PMID 28882127